CLINICAL TRIAL: NCT03419299
Title: Smart Phone/Device Application to Improve Delivery of Enteral Nutrition in Adult Patients Admitted to the Medical Intensive Care Unit
Brief Title: Smart Phone Application for Enteral Nutrition
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: OU 4496
Record Dates: First submitted 2018-01-13; First posted 2018-02-01 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Nutritional and Metabolic Diseases
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre- Application: Patients admitted prior to use of tube feeding application
- Post- Application: Patients admitted when tube feeding application was being used.
  Interventions: Other: Tube Feeding Application

INTERVENTIONS:
Other: Tube Feeding Application — A smart device application was developed and used to help residents determine the best enteral nutrition prescription for patients admitted to the ICU
  Groups: Post- Application

SUMMARY:
Internal medicine resident physicians were provided an ipod with the EN application to assist them in choosing EN formulas for patients during their ICU rotation. The primary outcome was improved initiation of EN within 24 hours of admission. Secondary outcomes include, time to initiate EN, goal calories reached, infections rates, length of stay, mortality, and concordance with clinical guidelines.

DETAILED DESCRIPTION:
Background: Resident physicians are frequently uncomfortable ordering enteral nutrition (EN) and are unaware of the variety of formulas and supplements available for different disease processes. Many depend on a clinical dietitian to assist with recommending EN formulas and patient energy requirements which may not be readily available upon patient admission. This creates a barrier to early initiation of EN and non-compliance with Society of Critical Care Medicine and American Society of Parenteral and Enteral Nutrition clinical guidelines. Objective: Internal medicine resident physicians were provided an ipod with the EN application to assist them in choosing EN formulas for patients during their ICU rotation. The primary outcome was improved initiation of EN within 24 hours of admission. Secondary outcomes include, time to initiate EN, goal calories reached. Design: This study is a retrospective chart review to evaluate the impact of a smart phone/device application (EN application) to assist resident physicians when ordering EN. The study is a single center trial conducted at an academic teaching facility. All patient data was obtained by a retrospective chart review of patients admitted to the intensive care unit (ICU) at The University of Oklahoma Medical Center.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the ICU
2. Require Mechanical Ventilation
3. Physician plans to order enteral nutrition for the patient

Exclusion Criteria:

1. Death likely within 24 hours
2. Needing parenteral nutrition
3. Cannot tolerate enteral nutrition for any reason

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical ICU patients who can tolerate enteral nutrition
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome was improved initiation of EN within 24 hours of admission | The time frame does involve a change in practice. The change is introduction of a smart app- 12 months prior to the smart device being used in the ICU by residents and 12 months during which the smart application was use by the ICU residents
  percent of patients with enteral nutrition ordered within 24 hours of admit compared to all patients admitted

SECONDARY OUTCOMES:
Total time to initiate EN | The time frame does involve a change in practice. The change is introduction of a smart app- 12 months prior to the smart device being used in the ICU by residents and 12 months during which the smart application was use by the ICU residents
  total hours between admit and when enteral nutrition is ordered
Percent of goal calories received prior to discharge from ICU | The time frame does involve a change in practice. The change is introduction of a smart app- 12 months prior to the smart device being used in the ICU by residents and 12 months during which the smart application was use by the ICU residents
  percent of calories received (a percent of the total recommended calories for the patient)

IPD SHARING:
Plan to Share IPD: No